CLINICAL TRIAL: NCT05723744
Title: Anonymized Data Collection From the CS6BP and Other Modalities for the Purpose of Developing Continuous Measurement of Heart Arrythmias
Brief Title: Anonymized Data Collection From the CS6BP for Heart Arrythmias Measurements
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CardiacSense Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CL00800
Record Dates: First submitted 2022-04-18; First posted 2023-02-13 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Heart Arrythmias
MeSH Terms: interventions — Electrocardiography, Ambulatory

STUDY DESIGN:
Intervention Model Description: The CS6BP includes a wrist-worn device with a clip connected to the band and is placed over the radial artery or a finger. The device includes a PPG sensor and is connected to ECG cables.
Masking Description: Open-label study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CS6BP , ECG holter and Blood pressure measurements (Experimental): The investigational device sensors tracings will be compared to the arrhythmia documented in all patients.
  Interventions: Device: ECG Holter and investigational device recordings for the purpose of developing Continuous Measurement of Heart Arrythmias

INTERVENTIONS:
Device: ECG Holter and investigational device recordings for the purpose of developing Continuous Measurement of Heart Arrythmias — For Candidates for pacemaker implantation: ECG Holter and investigational device recordings (of PPG, ECG, and motion sensors tracings non-invasively) will be recorded before procedure, during patient's hospitalization at cardiology division. Blood pressure values that are collected by an automated cuff will be collected including any notes attached to the values.
  All collected data will be analyzed offline

SUMMARY:
The purpose of this clinical study is to collect data simultaneously with the CS6BP watch sensors during EPS in order to characterize different evoked arrhythmias and record Blood Pressure during the procedures that blood pressure is collected by an automated cuff.

DETAILED DESCRIPTION:
The proposed clinical study is a Prospective Feasibility, Single-Center Study to collect data simultaneously with the CS6BP watch sensors during EPS or during admission in order to characterize different evoked arrhythmias. Subjects will be screened by the principal investigator or PI's delegate for meeting the study inclusion/exclusion criteria.

Subjects will be fitted with the CS6BP and ECG Holter by Investigator/Study Coordinator during the preparation of the subject to the procedure; when the subject is anesthetized and fitted with an automatic cuff that is preset to measure BP on a frequency as defined in the procedure protocol.

Subjects will be measured simultaneously with CardiacSense device, ECG Holter and EPS recording system if available (- ECG and intracardiac ECG recorded form intra-cardiac catheters). During the EPS the physician will timestamp and mark any provoked arrythmia either on ECG printouts or EPS recording system traces.

The device will be removed once patient has recovered. Subjects candidates for pacemaker implantation will be measured simultaneously with CardiacSense device and ECG Holter before procedure, during patient's hospitalization at cardiology division. At the end of the test the CardiacSense device and ECG Holter will be removed and their data will be downloaded. The recorded ECG (from Holter and if available also EPS recording/ mapping system) data will be analyzed by site staff. The analyzed ECG data will be sent to the company with the CS6BP raw data for further investigation.

BP values will be collected from subjects that are fitted with an automated cuff for BP monitoring for the purpose of evaluation and if required by the physician, during the hospitalization.

All adverse events (whether device related or not) will be reported during the course of the clinical study. All serious adverse events will be reported immediately to the study sponsor and monitor (within one working day). All clinical data will be recorded on appropriate CRFs.

ELIGIBILITY:
Inclusion Criteria:

* Age of eighteen (18) year and above
* In clinical need for electrophysiology study (standalone or before ablation procedure) and/or Subjects with AVB who are candidates for pacemaker implantation
* Ability and willingness to sign an informed consent form

Exclusion Criteria:

* Patients with significant co morbidities (assessed by the clinician at screening only):

Mechanically ventilated patients Mechanical circulation (LVAD, IABP, ECMO)

* Subjects who are currently enrolled in another clinical investigation in which the intervention might compromise the safety of the subject's participation in this study
* Subjects with PPG SNR <100 indicated by the CS6BP device
* Women who are pregnant or breastfeeding
* Subjects with had deformity banning from wearing the device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2020-11-27 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Data collection from the CS6BP watch sensors records , ECG holter and Blood pressure device for the purpose of developing Continuous Measurement of Heart Arrythmias | day 1, procedure day
  collection of data from the CS6BP sensors simultaneously with ECG Holter and EPS recorded signals to assess heart arrythmias present during EPS.

SECONDARY OUTCOMES:
Data collection from the CS6BP watch sensors records, ECG holter and blood pressure device for the purpose of developing Continuous Measurement of blood pressure | day 1, procedure day
  To collect data simultaneously with the CS6BP watch sensors during EPS in order to characterize different evoked Blood Pressure during the procedures that blood pressure is collected by an automated cuff.

CONTACTS AND LOCATIONS:
Overall Officials: Aharon Abbo, MD, Principal Investigator — Rambam Health Care Campus
Locations (1):
- Rambam Medical Center, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No